CLINICAL TRIAL: NCT04011111
Title: Objective and Subjective Evaluations of the Effect of Different Types of Intubation Tube Applications on Voice Performance in Early Postoperative Period
Brief Title: Intubation Tube Applications on Voice Performance in Early Postoperative Period
Status: Completed | Type: Observational
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Doğan Atan, Assoc. Prof., Hitit University
Other Study IDs: 2019/109
Record Dates: First submitted 2019-07-02; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Voice Alteration; Intubation Complication
Keywords: voice; intubation; subjective; objective
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Intubation tube and voice analysis — After the ıntubation tube application, done voice analysis early postoperative period

SUMMARY:
Changes in voice performance in the postoperative period due to trauma suffered during endotracheal intubation or edema occurring in the postoperative period are often observed. The present study aimed to evaluate the effect of different types of intubation tube applications on voice performance in the early postoperative period using objective and subjective voice analysis methods.

DETAILED DESCRIPTION:
A total of 88 patients who underwent endotracheal intubation either using a cuffed endotracheal (n = 44) or spiral-embedded cuffed endotracheal (n = 44) tube were included in this study. An endotracheal tube of 7.5 mm was used for female patients and that of 8 mm was used for male patients. A preoperative acoustic voice analysis was performed, and fundamental frequency (F0), jitter%, and shimmer% values were recorded. In addition, voice handicap index-30 (VHI-30) questionnaire was completed by the patients for subjective evaluation. The same procedure was repeated in the first 48 hours postoperatively. The preoperative and postoperative data were statistically compared. In addition, the effect of the type of endotracheal intubation tube on acoustic voice analysis parameters and VHI-30 scores was statistically evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years
* Conforming to the ASA I-II class according to the classification of the American Society of -Anesthesiologists (ASA)
* who were scheduled to undergo surgery that will not last more than 120 minutes

Exclusion Criteria:

* Patients with a lung disease
* Having obesity (BMI >35 kg.m-2)
* Pregnant patients
* Gastroesophageal reflux
* Suspected of having difficult airway (mouth opening <2.5 cm, Mallampati score >2, sternomental distance <12.5 cm, thyromental distance <6 cm, neck circumference >40 cm)
* A high risk of aspiration pneumonia
* Using inhaled steroids

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female adults
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
F0 (Fundemental frequency) | Preoperative period
  Acustic voice analysis parameter
Jitter% | Preoperative period
  Acustic voice analysis parameter
Shimmer% | Preoperative period
  Acustic voice analysis parameter
Voice Handicap Index-30 | Preoperative period
  Subjective voice analysis parameter

SECONDARY OUTCOMES:
F0 (Fundemental frequency) | Postoperative first 48 hours period
  Acustic voice analysis parameter
Jitter% | Postoperative first 48 hours period
  Acustic voice analysis parameter
Shimmer% | Postoperative first 48 hours period
  Acustic voice analysis parameter
Voice Handicap Index-30 | Postoperative first 48 hours period
  Subjective voice analysis parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University Faculty of Medicine, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No